CLINICAL TRIAL: NCT02423200
Title: A Randomized, Open-Label, Multiple Dose Clinical Pharmacology Study of Two Doses of a Selective p38 MAP Kinase Inhibitor, VX-745 in Patients With Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease (AD) or With Mild AD
Brief Title: Clinical Pharmacology of p38 MAP Kinase Inhibitor, VX-745, in Mild Cognitive Impairment Due to Alzheimer's Disease (AD) or Mild AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP14-745-303
Record Dates: First submitted 2015-04-03; First posted 2015-04-22 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — VX-745

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX-745 dose level 1 (Experimental): Active Group 1: VX-745 dose level 1 twice daily
  Interventions: Drug: VX-745
- VX-745 dose level 2 (Experimental): Active Group 1: VX-745 dose level 2 twice daily
  Interventions: Drug: VX-745

INTERVENTIONS:
Drug: VX-745 — Orally-active P38 MAP kinase alpha-selective inhibitor

SUMMARY:
This study will assess the effects of VX-745 on markers of disease in the central nervous system of patients with MCI due to AD or with mild AD. The study will also evaluate the safety and tolerability of VX-745 in these patients during 6 weeks of dosing, as well as the plasma and cerebrospinal fluid concentrations of VX-745 during dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 85 (inclusive)
* Willing and able to provide informed consent
* Clinical presentation consistent with MCI due to AD or of mild AD

  * Gradual progressive decline in memory function over >6 months
  * Amnestic presentation on neuropsychological testing with rapid forgetting (% reduction 1.5 standard deviations below the mean)
  * Clinical Dementia Rating (CDR) Sum of Box (SOB) score ≥0.5
  * Mini-Mental State Examination (MMSE) range: 20 to 30
* Brain hypometabolism by 18F-2-fluoro-2-deoxyglucose (FDG)-PET
* Participants may be taking medications for AD, provided that the dose of these medications has been stable for >3 months.

Exclusion Criteria:

* Evidence of neurodegenerative disease other than AD
* Inability for any reason to undergo MRI scans (e.g. pacemaker, vascular stent or stent graft). Patients who require sedation for screening procedures such as MRI may receive a short-acting sedative.
* Psychiatric disorder that would compromise ability to comply with study requirements
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
* Significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder or metabolic/endocrine disorders or other disease that would preclude treatment with p38 MAP kinase inhibitor and/or assessment of drug safety and efficacy
* Recent (<90 days) changes to AD medications prescribed for cognitive reasons or with the potential to impact cognition
* Psychotropic drugs taken within 1 month. Anticoagulant drugs taken within 1 week.
* Participation in a study of an investigational drug less than 6 months or 5 half-lives of the investigational drug, whichever is longer, before enrollment in the study
* Male subjects with female partner of child-bearing potential who are unwilling or unable to adhere to contraception requirements
* Female subjects who have not reached menopause or have not had a hysterectomy or bilateral oophorectomy/salpingoophorectomy
* Positive urine or serum pregnancy test or plans desires to become pregnant during the course of the trial
* Donation of >500 mL of blood or blood products within 2 months
* History of alcohol and/or illicit drug abuse within 6 months.
* Infection with hepatitis A, B or C or HIV.
* Any factor deemed by the investigator to be likely to interfere with study conduction

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hakop Gevorkyan, MD, Principal Investigator — Parexel
Locations (1):
- Parexel International, Glendale, California, United States

REFERENCES:
- [Derived] Tormahlen NM, Martorelli M, Kuhn A, Maier F, Guezguez J, Burnet M, Albrecht W, Laufer SA, Koch P. Design and Synthesis of Highly Selective Brain Penetrant p38alpha Mitogen-Activated Protein Kinase Inhibitors. J Med Chem. 2022 Jan 27;65(2):1225-1242. doi: 10.1021/acs.jmedchem.0c01773. Epub 2021 May 11. PMID 33974419

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the course of the study, and after one subject had been enrolled in the 125 mg dose group, FDA mandated the removal of the 125 mg dose group. As a result, the number subjects was revised downward to 9, 8 as planned in the 40 mg dose group and 1 in the 125 mg dose group.
Groups:
- Neflamapimod (VX-745) Dose Level 1: Active Group 1: VX-745 40 mg twice daily
  Neflamapimod (VX-745): Orally-active P38 MAP kinase alpha-selective inhibitor
- Neflamapimod (VX-745) Dose Level 2: Active Group 1: VX-745 125 mg twice daily
  Neflamapimod (VX-745): Orally-active P38 MAP kinase alpha-selective inhibitor
Period: Overall Study
Arm/Group | Neflamapimod (VX-745) Dose Level 1 | Neflamapimod (VX-745) Dose Level 2
Started | 8 | 1
Completed | 7 | 1
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VX-745 Dose Level 1 | VX-745 Dose Level 2 | Total
Number analyzed (Participants) | 8 | 1 | 9
Age, Continuous [Median (Full Range); unit: years] | 71 [66 to 74] | 68 [68 to 68] | 71 [66 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: count of participants]
  United States | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to End of Treatment in Cerebrospinal Fluid Levels of Cytokines
Description: Cytokines: Of nine cytokines assessed, only CSF IL-8 quantifiable at all time points. And so, only IL-8 levels are being reported herein. The analysis was exploratory and no statistical analysis was performed.
Time Frame: Baseline and Day 42 of dosing with VX-745
Population: As there was only one subject in the 125 mg dose group (see Pre-Assignment Details), and the blood concentration levels in this subject was similar to that in 125 mg dose group, this subjects data was combined with the 40 mg dose group in this analysis. In addition, two subjects did not have Day 42 CSF samples available for analysis
Measure: Mean (Standard Deviation); unit: percentage of baseline at Day 42
Groups:
- Overall Study Population: Combined 40 mg and 125 mg subjects; N=7 with baseline and Day 42 results
Arm/Group | Overall Study Population
Number analyzed (Participants) | 7
percentage of baseline at Day 42 | 137 (115)

2. Secondary Outcome: Severe or Serious Adverse Events
Description: Number of patients with severe or serious adverse events
Time Frame: At baseline and at each study visit during (days 1, 7, 14, 21, 28, 35 and 42) and after (day 51) dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Neflamapimod (VX-745) Dose Level 1 | Neflamapimod (VX-745) Dose Level 2
Number analyzed (Participants) | 8 | 1
Participants | 0 | 0

3. Secondary Outcome: Maximal CSF VX-745 Concentration
Description: Ratio fo CSF to plasma drug concentration at time matched time points. Samples taken
Time Frame: All samples with quantifiable CSF drug levels were included (n=12). Eight were obtained 3-hours post-dose, either on Day 1 (n=4) or Day 42 (n=4). 3 samples were at 6-hours post-dose on Day 42; and one was at 6-hours post-dose on Day 1.
Population: As there was only one subject in the 125 mg dose group (see Pre-Assignment Details), and the blood concentration levels in this subject was similar to that in 125 mg dose group, this subjects data was combined with the 40 mg dose group in this analysis.
Measure: Mean (Standard Deviation); unit: ratio of plasma drug concentration
Groups:
- Overall Study Population: Combined 40 mg and 125 mg subjects
Arm/Group | Overall Study Population
Number analyzed (Participants) | 9
ratio of plasma drug concentration | 0.062 (0.01)

4. Secondary Outcome: Episodic Memory Function
Description: Total Recall in Hopkins Verbal Learning Test (HVLT). Range is 0-36, with increases in score indicating improvement in cognitive function.
Time Frame: Change from baseline to Day 42
Population: As there was only one subject in the 125 mg dose group (see Pre-Assignment Details), and the blood concentration levels in this subject was similar to that in 125 mg dose group, this subjects data was combined with the 40 mg dose group in all outcome measure analyses. In addition, one subject did not have a Day 42 HVLT-R analysis.
Measure: Mean (Standard Deviation); unit: points on HLVT Total Recall (range 0-36)
Arm/Group | Overall Study Population
Number analyzed (Participants) | 8
points on HLVT Total Recall (range 0-36) | 3.5 (3.6)

ADVERSE EVENTS:
Groups:
- Overall Study Population: Combined 40 mg and 125 mg subjects. As there was only one subject in the 125 mg dose group (see Pre-Assignment Details), and the blood concentration levels in this subject was similar to that in 125 mg dose group, this subjects data was combined with the 40 mg dose group in the adverse event analysis.
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Population (N=9)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical study was conducted at at clinical pharmacology unit owned by a contract research organization (CRO; Parexel) that was contracted by the sponsor to conduct the study. Site principal investigator is an employee of a contract research organization. As per the contract, the sponsor has "all rights, title and interest in the results".